CLINICAL TRIAL: NCT04602182
Title: EFFECTS OF AN INTERVENTION WITH MUSICOTHERAPY IN THE WEANING FROM MECHANICAL VENTILATION IN PATIENTS OF THE INTENSIVE MEDICINE UNIT OF THE ALAVA UNIVERSITY HOSPITAL
Brief Title: Effectiveness of Musicotherapy in Weaning From Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Collaborators: AGRUPARTE S.L. (Unknown)
Responsible Party: Principal Investigator, Esther Corral Lozano, intensive medicine physician, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MusicoT
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Weaning; Respiration, Artificial; Music Therapy
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Single-blind randomized clinical trial in parallel groups and controlled with standard clinical practice.
Who Masked: Outcomes Assessor
Masking Description: The person responsable for carrying out the statistical analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy gruop (experimental group) (Experimental): Experimental group: Patients will receive a daily music therapy intervention from the beginning until the end of the weaning from mechical ventilation.
  Interventions: Procedure: music therapy intervention
- control group (Active Comparator): Control group: Patient will follow the usual clinical practice for the weaning from mecanichal ventilation to the end of the weaning.
  Interventions: Procedure: music therapy intervention

INTERVENTIONS:
Procedure: music therapy intervention — Patients will receive a daily music therapy intervention from the beginning until the end of the weaning from mechical ventilation.

SUMMARY:
1. OBJECTIVES:

   General objective: Assess the effects of a music therapy intervention during the weaning from the mechanical ventilation in a group of patients, and compare it to the usual clinical practice.

   Specific objectives: Main objective: assess the effect of a music therapy intervention on the length of the weaning in a group of critical patients, and compare it to a group of critical patients who receive the usual clinical practice.

   Secondary objectives:
   * Compare the levels of sedo-analgesia required in critical patients receiving the music therapy intervention during the process of weaning versus the levels of sedo-analgesia required by the control group.
   * Compare the Anxiety-agitation level in critical patients receiving the music therapy intervention during the process of weaning, versus the anxiety-agitation leved felt by the control group.
   * Compare the level of pain in critical patients receiving the music therapy intervention during the weaning versus the level of the pain felt by the control group.
   * Compare the level of delirium in critical patients receiving music therapy during the weaning versus the level of delirium of the control group.
   * Compare heart and breath frequency, blood pressure and oxygen saturation in critical patients receiving music therapy during the mechanical ventilation extubation (weaning) process, versus the index of control group.
   * Compare the stress perceived in critical patients receiving music therapy intervention during the mechanical extubation process, versus the level of the control group, which receives the usual medical care (without intervention with music therapy), 90 days after Inico of the process, Perceived the Stress Scale (PSS).
   * Describe and analyze the experience by the patient of the intervention with music therapy the weaning process and the coping strategies possible for musicotherapeutic intervention, using a Semi-instructed interview that takes place at 90 days beginning the process.
2. DESIGN: single blind clinical trial in parallel groups, single blind clinical trial.
3. POPULATION of this study are patients who initiate weaning for ventilation mechanics.

DETAILED DESCRIPTION:
Experimental group: Patients will receive a daily music therapy intervention from the beginning until the end of the weaning from mechical ventilation.

Control group: Patient will follow the usual clinical practice for the weaning from mecanichal ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation for at least 48 hours, with the decision to start the process of weaning, which comes determined by the decision to switch from controlled mode to support or spontaneous breathing modalities.

Exclusion Criteria:

* Patients with established moderate-severe psychiatric pathology.
* Patients with severe hearing deficit.
* Patients in whom the Limitation of Life Support Treatment (LTSV) has been decided and have a life expectancy of less than 48h.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-06-19 (Estimated)

PRIMARY OUTCOMES:
Lenght of weaning from mechanical ventilation (hours) | within 1 week
  Time in hours from the beginning to the end of the disconnection process

SECONDARY OUTCOMES:
Sedoanalgesia average dosis | within 1 week (during the weaning)
Score on the Richmond Agitation scale-24 hours prior to the start of the study, and every eight hours during the study and at the end of the mechanic ventilation disconnection period | within 1 week (during the weaning)
  RASS scoring and interpretation should be based on the sedation protocol being used. For minimal sedation protocols (RASS -2 to 0), sedation should be modified or decreased for a RASS score of -3 or less.[3] Scores of 2 to 4 may indicate under-sedation. At minimum, the patient should be assessed for pain, delirium, and anxiety. In addition, other underlying causes of agitation should be investigated and treated as appropriate.
  In select cases, a deep sedation protocol (RASS -4 and -5) may be used.[3] For scores of -3 or higher, sedation should be modified to achieve the desired range
Score on the Confusion Assessment Method scale for Intensive Care Units (CAM-ICU) 24 hours prior to the start of the study, and every eight hours during the study and at the end of the mechanical ventilation disconnection period | within 1 week (during the weaning)
  Rate each symptom of delirium listed in the instrument as absent (0), mild (1), or marked (2), except acute onset or fluctuating course which was rated as absent (0) or present (1). The severity score is created by an additive summary of the ratings ranging from 0-7 (short form) and 0-19 (long form). Higher scores indicate more severe delirium.
Systolic TA (mm hg) at the beginning, at the end of the intervention, and 30 minutes after the end | within 1 week (during the weaning)
Diastolic TA (mm hg) at the beginning, at the end of the operation, and 30 minutes after the end | within 1 week (during the weaning)
Heart rate (beats/minutes) at the beginning, at the end of the intervention, and 30 minutes after the end | within 1 week (during the weaning)
Breathing frequency at the beginning, at the end of the speech, and 30 minutes after the end | within 1 week (during the weaning)
Oxygen saturation, at the beginning, at the end of the intervention, and 30 minutes after the end | within 1 week (during the weaning)
Perceived Stress Scale (PSS) score | 90 days after the start of the weaning process
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceivedstress. ►Scores ranging from 0-13 would be considered low stress. ►Scores ranging from 14-26 would be considered moderate stress.►Scores ranging from 27-40 would be considered high perceived stress.
Perception of the influence of the Music Therapy Intervention and intervention strategies, through a Semi-structured Interview | 90 days after having started the process of disconnecting the mechanical ventilation (weaning)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Araba university hospital, Vitoria-Gasteiz, Alava
  - Esther Corral, Vitoria-Gasteiz, Alava